CLINICAL TRIAL: NCT00159094
Title: A Phase II Trial of Doxil and Multiday Vinorelbine in Patients With Metastatic Breast Cancer
Brief Title: A Trial of Doxil and Multiday Vinorelbine in Patients With Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hematology Oncology Consultants (Other)
Collaborators: Ortho Biotech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO03-21-005
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2008-06-02 (Estimated); Status verified 2005-09

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Vinorelbine

INTERVENTIONS:
Drug: Doxil and Vinorelbine

SUMMARY:
This is a phase II trial of Doxil on day 1 and vinorelbine on days 1 and 2 in women with metastatic breast cancer. Administered every 28 days. A study to assess the safety and efficacy of Doxil and vinorelbine in metastatic breast cancer.

DETAILED DESCRIPTION:
PROTOCOL SUMMARY

Study design: Phase II trial of monthly Doxil® and vinorelbine on day 1 and 2 in women with metastatic breast cancer.

Treatment plan: Patients will continue therapy, until they have unacceptable toxicity or disease progression.

Primary endpoint: Response rate

Secondary endpoints: Time to progression, overall survival and toxicity.

Additional study objectives: Evaluation of treatment-related dyspnea, with measurement of pulse oximetry during and after drug administration, and rigorous study of patients who experience dyspnea. Palmar-plantar erythrodysesthesia (PPE) will be treated with one of 2 randomly assigned topical salves, measuring duration and severity of symptoms.

Eligibility: Women who have had prior chemotherapy in the adjuvant or metastatic setting, or both, up to 3 prior regimens. Patients having more than one prior regimen for metastatic disease must have a performance status of 0 or 1; others may have 0-2. No prior Doxil® or vinorelbine therapy. Patients are ineligible if prior anthracycline dose is greater than 400 mg/m2, or if they have primary anthracycline-refractory disease, with disease progression during treatment or with relapse/recurrence within 6 months after last dose of anthracycline. Patients must have normal neurologic, hematologic, renal and hepatic functional parameters. Asymptomatic brain metastases are permissible.

Treatment plan: Doxil® 40 mg/m2 IV infusion over 60 minutes on day 1 Vinorelbine 15 mg/m2 IV over 6 minutes on days 1 and 2 Dexamethasone 4 mg IV or 8 mg po (Doxil® pretreatment) Heparin 5000 U IV (Vinorelbine pretreatment) Pyridoxine (vitamin B6) 200 mg po qd Repeat every 28 days.

Supportive measures:

For anemia (hematocrit < 35): Procrit® 40,000 U q wk For neutropenia (ANC < 1,000/mm3 ): Prophylactic antibiotics (Cipro® or Septra®) For all cycles after neutropenic fever/infection or grade 3-4 stomatitis: Prophylactic Neulasta® 6 mg SQ on day 3 (This intervention may be adopted for all patients, all cycles, if 2 of the first 4 patients enrolled need it.) For PPE: randomize between 2 topical salves and document duration and severity of sx

Dose adjustments: Subsequent cycles are given on day 29 or after recovery or to grade 0-1 toxicity, with no more than 3 weeks delay. Reduce dose of both drugs by 25% if grade 3 or 4 stomatitis or palmar-plantar or grade 4 thrombocytopenia. Reduce dose of Doxil® ONLY by 50-75% if abnormal bilirubin, alkaline phosphatase and/or ALT, AST (appendix 14.3)

ELIGIBILITY:
Inclusion Criteria:

* Patients must be informed of the investigational nature of this study and must give and sign informed consent in compliance with federal and institutional guidelines.
* Women 18 years or older with biopsy proven advanced breast cancer.
* Patients with reproductive potential must use an adequate contraceptive method (e.g., abstinence, intrauterine device, oral contraceptives, barrier device with spermicide, or surgical sterilization) during treatment and for three months after completing treatment.
* Performance status (PS) 0-2 (ECOG). PS must be 0-1 if patient has had more than one prior regimen for metastatic disease or more than 2 prior regimens, including adjuvant and metastatic.
* Measurable disease by RECIST criteria, with baseline staging completed within 14 days of registration.
* At least two weeks post surgery and three weeks from completion of irradiation and recovered from toxicities associated with these treatments.
* Psychological, family, social and geographical conditions allowing weekly medical follow up during chemotherapy are required.
* Preregistration blood work must include complete blood counts with differential, and blood chemistries including serum bilirubin, GGT, LDH, SGOT, SGPT, alkaline phosphatase, creatinine, and tumor markers, CEA and CA 27-29. Patients must have:

  * Absolute neutrophil count (ANC) >1,500/mm3
  * Platelet count >100,000/mm3
  * Hemoglobin > 8.0 g/dl
  * Serum creatinine < 2.5 mg/dl (< 200 mol/L)
  * Serum bilirubin < the upper limit of normal (ULN)
  * SGOT and SGPT or AST and ALT < 2.0 x ULN
  * Alkaline phosphatase < 2.0 x ULN, except if attributed to tumor
  * Life expectancy > than 12 week.

Exclusion Criteria:

* Prior Doxil® or vinorelbine
* Cumulative anthracycline dose exceeding 400 mg/m2 anthracycline
* Primary anthracycline refractory disease, ie. disease progression during treatment or relapse/recurrence within 6 months after last dose of anthracycline
* If PS 0-1, more than 3 prior chemotherapy regimens, including adjuvant and metastatic
* If PS 2, more than 1 prior regimen for metastatic disease or more than 2 prior chemotherapy regimens, including adjuvant and metastatic
* Hormone therapy including aromatase inhibitors within 2 weeks of baseline
* Pregnant or lactating women. Women of reproductive potential must have a negative pregnancy test and must agree to use an effective contraceptive method
* Prior history of cardiac disease, with New York Heart Association Class II or greater, or clinical evidence of congestive heart failure
* Symptomatic brain metastasis
* Past medical history of severe hypersensitivity reaction to conventional formulation of doxorubicin HCL or the components of Doxil® or vinorelbine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-10

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
Time to progression
Overall survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Leslie R Laufman, MD, Principal Investigator — Hematology Oncology Consultants, Inc
Locations (2):
- United States (2):
  - Hematology Oncology Consultants, Inc, Columbus, Ohio
  - Hematology Oncology Consultants, Inc, Newark, Ohio